CLINICAL TRIAL: NCT04354116
Title: Microimplant-assisted Rapid Palatal Expansion Appliance to Orthopedically Correct Midface Deficiency in Patients With Cleft Lip and Palate: a Randomized Clinical Trial
Brief Title: MARPE in Patients With Cleft Lip and Palate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontifícia Universidade Católica de Minas Gerais (Other)
Responsible Party: Principal Investigator, Ildeu Andrade Jr., Principal Investigator, Pontifícia Universidade Católica de Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MARPE Class III cleft patients
Record Dates: First submitted 2020-04-01; First posted 2020-04-21 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Palatal Expansion Technique; Cleft Lip and Palate; Class III Malocclusion; Skeletal Malocclusion
Keywords: palatal expansion technique; Cleft Lip; Cleft Palate; Maxillary retroposition
MeSH Terms: conditions — Cleft Lip; Malocclusion, Angle Class III; Cleft Palate; Retrognathia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MARPE (Experimental): Maxillary expander anchored in mini-implants (MARPE)
  Interventions: Device: Rapid maxillary expansion; Device: Maxillary Protraction
- Hyrax (Active Comparator): Tooth-born anchored maxillary expanders, without mini-implants
  Interventions: Device: Rapid maxillary expansion; Device: Maxillary Protraction

INTERVENTIONS:
Device: Rapid maxillary expansion — Palatal expanders of the HYRAX type, with bands on the first permanent molars will be used for patients in both groups. In the experimental group, the expander will be anchored mesially and bilaterally in mini-implants, in a technique known as rapid maxillary expansion assisted by mini-implants (MARPE). The control active group will be with conventional HYRAX expanders. The maxillary expansion protocol will be once a day for 2 weeks.
Device: Maxillary Protraction — Protraction hooks will be projected around the upper canine area. In the experimental group (MARPE), the appliance will be anchored mesially and bilaterally in mini-implants. The control active group will be anchored with conventional HYRAX expanders. Both groups will be treated with maxillary protraction with a Petit-type face mask at night (12 hours a day).

SUMMARY:
The objective of this randomized controlled study will be to evaluate the dental and skeletal effects of maxillary protraction with a facemask, associated with MARPE and Class III elastics in patients with unilateral cleft lip and palate (CLP) with maxillary retrusion, compared to HYRAX type maxillary expanders. The investigators will examine differences in treatment times, along with skeletal, dental and soft tissue changes.

DETAILED DESCRIPTION:
The CONSORT statement will be used as a guide for this study. This work will be a parallel group study, randomized, with active control, with an allocation ratio of 1: 1.

This study was submitted to the Research Ethics Committee of the Pontifical Catholic University of Minas Gerais. Participants will be recruited in the Master's Degree in Orthodontics at PUC Minas, based on inclusion criteria.

Interventions:

Palatal expanders of the HYRAX type, with bands on the first permanent molars or second deciduous molars will be used for patients in both groups. The hooks for the use of Class III elastics will be welded on the vestibular of the upper molar bands. In the experimental group, the expander will be anchored mesially and bilaterally in mini-implants, in a technique known as rapid maxillary expansion assisted by mini-implants (MARPE). The control group will be active, with conventional dento-mucus-supported HYRAX expanders. All expanders will be manufactured by the same orthodontic technician.

Both groups will be treated with maxillary protraction with a Petit-type face mask at night (12 hours a day). The direction of the elastics for the maxillary traction force will be between 15˚ to 30˚ below the occlusal plane, providing a force between 400 and 500 g per side. During the day (12 hours a day), patients will use a lower expansion plate with an occlusal stop, which will be activated once a week (0.25 mm), with hooks in the region of the lower canines for the use of Class III elastics. size 3/16 "(150g). The time-frame of the experiment will be 6 months.

Results (primary and secondary) The primary outcome will be the degree of anterior movement of the maxilla after treatment). Secondary outcomes will be changes in other cephalometric variables and treatment time.

Conical beam computed tomography (CBCT) will be performed at the beginning and at the end of the treatment. Teleradiographies will be extracted from the CFFCs and cephalometric measurements will be obtained by the investigator (V.E.) using the Dolphin Image software (Austin, USA). Traditional cephalometric measurements will be used to describe the changes before and after treatment.

Calculation of the sample size As no study in the orthodontic literature used the same protocol used in this study, the sample size will be estimated by G * Power (version 3.0.8), with 95% power; significance level of 5%; two-tailed. For point A, sagittal movements of 2.6 +/- 1.5 mm in the RME group and 5.8 +/- 2.3 mm in the RME group with constriction, a minimum sample size of 11 in each group will be necessary to detect a significant difference between groups. For ANS, sagittal movements of 2.1 +/- 1.3 mm in the RME group and 4.8 +/- 2.5 mm in the RME group with constriction, a minimum sample size of 16 in each group will be necessary to detect a significant difference between groups. Therefore, 16 will be the minimum sample size for each group. The sample size will be increased by 40%, resulting in 22 patients for each group, in case there is a withdrawal or the need to use a different protocol.

Randomization (random number generation, allocation hiding, implementation) Patients will be recruited and allocated to the control group (RME) or the intervention group (MARPE) according to the sequence of participation. Simple randomization will be applied.

Blinding The blinding of investigators or participants will not be possible because the expanders in the two groups will be different. Operators and patients will easily know which group they are in. However, blinding will be used during cephalometric analysis. All image exams will be hidden by opaque tape and replaced with research numbers and then mixed together before analysis. The investigator will not know the clustering of the CT scans, which will look similar.

Statistical analysis (primary and secondary results, subgroup analyzes) All statistical analyzes will be performed using the software (version 18.0; PASW Statistics, Chicago, Illinois). Descriptive statistics will include the means and standard deviations of age, total treatment time, maxillary prostration time, cephalometric values and changes in values in each group. The 1-sample Kolmogorov-Smirnov test will be used to test the normality of distributions for all times and differences in cephalometric values. Independent t-tests will be used to compare the two groups, including total treatment time, protraction time and changes in cephalometric values; the t-tests will be used for the values that show "equality of variances not assumed" between the groups (SNA and Nasio perpendicular). The level of significance will be 0.05, with two-tailed test.

Error of the Method All locations and measurements of the points will be checked twice carefully at the end of the initial plots and measurements. Not all images will be traced twice. However, to evaluate the tracing errors, 20 scans will be chosen at random. Plots, locations and measurements will be made twice, two weeks apart and then subjected to the Dahlberg formula. The error of the method will be determined by the Dahlberg formula, where n = 20 and d will be the difference between the measurements in 2 moments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cleft lip and palate;
* 6 to 13 years before orthodontic treatment, with sagittal deficiency of the facial middle third;
* Angle Class III malocclusion, or mesial step of the deciduous second molars, and anterior crossbite;
* ANB less than 0˚, Wits less than -2 mm and the distance from point A to the perpendicular nasion less than 0 mm.

Exclusion Criteria:

* Previous orthodontic treatment;
* Other craniofacial anomalies;
* Inadequate maxillary denture for placement of a expander.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-09-10 (Estimated); Study Completion 2021-09-10 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the degree of anterior movement of the maxilla after treatment). | 6 months
  Cone beam computed tomography (CBCT) will be performed at the beginning and at the end of the treatment. Three-dimensional virtual models, built from the CBCT's scans, will allow to measure the changes between T0 and T1. The processing of the TCFC and virtual models will be done using the ITK-SNAP 2.2 software (free software, www.itksnap.org), SLICER CMF 4.0 (free software, www.slicer.org).

SECONDARY OUTCOMES:
Secondary outcomes will be changes in other cephalometric variables and treatment time. | 6 months
  Cone beam computed tomography will be performed at the beginning and at the end of the treatment. Three-dimensional virtual models, built from the CBCT's scans, will allow to measure the changes between T0 and T1. The processing of the TCFC and virtual models will be done using the ITK-SNAP 2.2 software (free software, www.itksnap.org), SLICER CMF 4.0 (free software, www.slicer.org).

CONTACTS AND LOCATIONS:
Overall Officials: Ildeu Andrade Jr., PhD, Principal Investigator — Pontifícia Universidade Católica de Minas Gerais
Locations (1):
- Pontifical Catholic University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No